CLINICAL TRIAL: NCT06082973
Title: Evaluation of Dual-hormone Artificial Pancreas With Closed-loop Glucose Control Versus Single-hormone With Carbohydrate Recommendations Under Unannounced Exercise and Meal Challenge in Adults With Type 1 Diabetes.
Brief Title: Dual-hormone Artificial Pancreas Versus Single-hormone Under Exercise and a Meal Challenge
Acronym: TAILOR/3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de València (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Jorge Bondia, Jorge Bondia Company, Universitat Politècnica de València
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAILOR/3
Record Dates: First submitted 2023-09-05; First posted 2023-10-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: artificial pancreas; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: Device: closed-loop control algorithm with a dual-hormone configuration versus a single-hormone configuration with rescue carbohydrate recommendations for glucose control during an unannounced 30-min aerobic exercise session and a meal challenge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-hormone configuration system (insulin and glucagon) (Experimental): 12-hour inpatient study that will include an unannounced 30-min aerobic exercise session and a meal challenge. Automated insulin and glucagon delivery will be performed using a dual-hormone configuration system for glucose control .
  Interventions: Device: Automated insulin delivery system algorithm with a dual-hormone configuration (insulin and glucagon) for glucose control
- Single-hormone configuration (insulin) with carbohydrate recommendations system (Active Comparator): 12-hour inpatient study that will include an unannounced 30-min aerobic exercise session and a meal challenge. Automated insulin delivery will be performed using a single-hormone configuration system with carbohydrate recommendations if needed for glucose control .
  Interventions: Device: Automated insulin delivery system with a single-hormone configuration (insulin) with rescue carbohydrate recommendations for glucose control

INTERVENTIONS:
Device: Automated insulin delivery system algorithm with a dual-hormone configuration (insulin and glucagon) for glucose control — Participants will wear a CSII system with the CGM device. Insulin will be administered through the AID dHmG system, and microdoses of glucagon (GlucaGen®) will be subcutaneously administered based on automatic recommendations for hypoglycemia mitigation. The subcutaneous administration of reconstituted glucagon will be conducted using a 0.5 mL insulin syringe with needle, allowing for precise doses as small as 0.01mg/0.01 mL.
  Other Names: Dual-hormone configuration system controller
  Arms: Dual-hormone configuration system (insulin and glucagon)
Device: Automated insulin delivery system with a single-hormone configuration (insulin) with rescue carbohydrate recommendations for glucose control — Participants will wear a CSII system with the CGM device. Insulin will be administered through the AID sHC system, along with automatic rescue carbohydrate recommendations for hypoglycemia mitigation. As per the carbohydrate recommendation, participants will received the suggested amount of carbohydrates using an oral glucose gel containing 15g of carbohydrates per unit.
  Other Names: Single-hormone configuration system with rescue carbohydrate recommendations controller
  Arms: Single-hormone configuration (insulin) with carbohydrate recommendations system

SUMMARY:
The present clinical trial aims to examine alternative strategies for preventing/mitigating hypoglycemic events among adults with type 1 diabetes utilizing a highly personalized control system. This system offers two configurable options: a single-hormone configuration with automatic rescue carbohydrate recommendations (sHC) and a dual-hormone configuration with subcutaneously administered glucagon boluses (dHmG). The main question addressed in this study focuses on determining whether the dHmG outperforms the sHC in terms of minimizing the time spent below the target range and number of hypoglycemic events.

Each participant will undergo two 12-hour controlled inpatient studies, including each an unannounced 30-min aerobic exercise session and a meal challenge. The order of these studies, comparing the dHmG to the sHC, will be randomized.

DETAILED DESCRIPTION:
RATIONALE OF THE STUDY

Automated insulin delivery (AID), commonly referred to as artificial pancreas, represents the most advanced treatment for individuals with type 1 diabetes (T1D). AID is recognized for its ability to optimize insulin treatment, thereby maximizing the time spent within the target range (TIR) while minimizing instances of blood glucose levels falling below or exceeding the target range. At present, several hybrid AID systems are commercially available, primarily in the EU and US, providing this population with the benefits of this advanced therapy. Despite the benefits offered by current AID systems and diabetes technology in general for the treatment of T1D, only approximately 20% of individuals achieve the recommended glycemic target. The existing systems heavily rely on timely and accurate information from the user regarding two significant glycemic disturbances: meals and physical activity. Overestimation of carbohydrate intake and physical activity are the primary drivers contributing to postprandial and episodic hypoglycemia, respectively, with potential consequences during the overnight period.

The current investigation aims to examine alternative strategies for preventing/mitigating hypoglycemic events utilizing a highly personalized control system. This system offers two configurable options: a single-hormone configuration with automatic rescue carbohydrate recommendations and a dual-hormone configuration with subcutaneously administered glucagon boluses. The research question addressed in this study focuses on determining whether the dual-hormone configuration outperforms the single-hormone with rescue carbohydrate recommendations configuration in terms of minimizing the time spent below the target range.

HYPOTHESIS

Our hypothesis suggests that the utilization of the dual-hormone configuration will result in a decrease in the amount of time spent below the target range (70-180 mg/dL) and a reduction in the number of hypoglycemic events in comparison to the single- hormone configuration with automatic rescue carbohydrate recommendations.

MAIN OBJECTIVES

Primary objectives of this study are: (1) to evaluate the duration of time spent below the target range (70-180 mg/dL) and (2) to assess the occurrence of Level 1 (<70 mg/dL) and Level 2 (<54 mg/dL) hypoglycemic events. These objectives will be examined within the context of a 12-hour, highly supervised, controlled, randomized clinical trial that incorporates real-life challenges. These challenges will involve an unannounced 30-min aerobic exercise session, as well as the consumption of a meal that will be announced.

INVESTIGATIONAL PLAN

Study design:

This study follows a longitudinal, prospective, randomized crossover interventional design. Each participant will undergo two inpatient studies, including an unannounced exercise session and a meal challenge. The order of these studies, comparing the dual-hormone configuration (dHmG) to the single-hormone configuration with rescue carbohydrate recommendations (sHC), will be randomized. The study will comprise five visits:

Visit 1: Screening visit. This visit will take place one week prior to Visit 2. During the screening visit, patients will provide informed consent, undergo examinations, and undergo tests to ensure their safety in participating in the study. Each subject will also be instructed to wear a continuous glucose monitoring (CGM) device.

Visit 2: Randomization visit an Incremental Exercise test. This visit will take place 2 weeks before Visit 3. Patients will be assigned to one of two randomization schedules and will receive further instructions regarding their participation in the study. All necessary materials for conducting CGM will be provided during this visit. Additionally, an incremental exercise test will be conducted during this visit to determine the optimal intensity for the aerobic exercise sessions.

Visits 3 and 4: Experimental study days. Each subject will undergo two interventions, consisting of an unannounced 30-min aerobic exercise test and a 60 g carbohydrate meal challenge. These interventions will occur at 2-3 week intervals (wash-out period), allowing for the completion of the two experiments within approximately 3 weeks.

Visit 5: Final visit (follow-up visit). This visit will take place 1 week after the conclusion of Visit 4. Subjects will undergo a physical examination, and safety variables will be determined in the laboratory, following the same procedures outlined in Visit 1.

Study population:

Fifteen adults, ranging in age from 18 to 65 years, who have been diagnosed with T1D for more than 1 year and do not have advanced chronic micro- and macroangiopathic diabetic complications, will be recruited from individuals attending the Diabetes Unit at the Hospital Clínico Universitario de Valencia. These individuals must be on intensive insulin treatment with continuous subcutaneous insulin infusion (CSII) and have fair metabolic control (HbA1c <9.0%) while not experiencing hypoglycemia unawareness. Out of the recruited participants, five individuals will undergo an initial feasibility test for the dual-hormone (dHmG) configuration, while, subsequently, ten individuals will be randomly assigned to the dHmG vs. sHC study.

Sample size:

Five adults with T1D will initially participate in a preliminary feasibility study testing the dHmG. Subsequently, an additional ten adults with T1D will be enrolled in the interventional study comparing dHmG versus sHC. As the present study is exploratory in nature, a formal determination of the sample size was not calculated.

Study procedure and schedule:

The study will commence with a preliminary stage focused on evaluating the safety and feasibility of the coordinated dHmG (consisting of AID with manual glucagon administration) in five adults diagnosed with T1D. Following confirmation of safety data by the data and safety monitoring board, ten adult participants will be randomly assigned to the order in which the modalities (dHmG and sHC) will be tested, following a brief algorithm refinement procedure.

Description of study days:

Visit 1 (screening visit): After patients have provided informed consent, a series of examinations and tests will be conducted a week prior to Visit 2, including: Medical History, Physical examination, Standard 12-lead ECG, Clinical Laboratory Tests, detection of asymptomatic hypoglycemia using a validated Spanish version of the Clarke Test questionnaire, short version of the International Physical Activity Questionnaire to all participants and metabolic equivalents (METS) calculation.

Visit 2 (randomization visit and incremental exercise test): If the outcome of the first visit is favorable, patients will be eligible for enrollment in the study and undergo randomization. They will be provided with instructions on the use of CGM for two weeks of monitoring prior to the commencement of the experimental study visits, which includes system calibration and preparation. Additionally, an incremental exercise test will be conducted during this visit to determine the optimal intensity for the aerobic exercise sessions.

Visits 3 and 4 (intervention days): Each subject will undergo two study sessions, each of which will include an unannounced aerobic exercise test and a 60 g carbohydrate meal challenge that will be announced. The algorithm will utilize the individual's insulin/carbohydrate ratio to calculate the meal insulin bolus without any reduction. These sessions will be scheduled at intervals of 2-3 weeks and assigned randomly. In one session, the dHmG configuration for glucose control will be employed, while the sHC will be used in the other session. Participants will wear a CSII system with the CGM device.

Visit 5 (follow-up visit): Subjects will be required to attend a follow-up visit after completing the two study days. During this visit, a physical examination and laboratory safety variables, as described in Visit 1, will be repeated.

Study duration:

The anticipated duration of this study will be four months, with subject recruitment scheduled to commence in December 2023 and the completion of experiments projected for March 2024.

ETHICAL AND LEGAL ASPECTS

The procedures set out in this study protocol, pertaining to the conduct, evaluation, and documentation of this study, are designed to ensure that the sponsor and investigator (in this case the same person) comply with the principle of the good clinical practice guidelines and the Declaration of Helsinki in the conduct, evaluation and documentation of this study. The study will also be carried out in keeping with local legal requirements.

This study involves the collection and use of biological samples for research purposes, in accordance with the provisions of Law 14/2007 on biomedical research and Royal Decree 1716/2011 on Biobanks.

An informed consent document that includes both information about the study and the consent form will be prepared and given to the subjects. The documents will be in a language understandable to the subject and will specify who will inform the subject.

The study database will not contain any information that could allow the individual identification of the study participants. The data obtained will be used exclusively for the purposes described in this research project. The information will be treated as confidential and will be stored and processed in accordance with the provisions of European Union (EU) Regulation 2016/679 of the European Parliament and the Council of 27 April 2016 on the protection of personal data and the free movement of such data, as well as Organic Law 3/2018 of December.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* CSII treatment for a minimum of 6 months prior to Visit 1.
* Body mass index between 18 and 30 kg/m2.
* HbA1c level below 9.0% at Visit 1.
* Physical examination, laboratory data, and ECG (electrocardiogram) results are within normal limits. Clinically insignificant abnormalities, as determined by the investigator, will not be considered exclusion criteria.
* Postmenopausal women or women of childbearing age who have a negative urine pregnancy test during the screening visit.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Hypoglycemia unawareness (as indicated by a Clarke Test score greater than 3).
* Presence of progressive, fatal disease.
* History of drug or alcohol abuse.
* History of being HIV positive, active hepatitis B or hepatitis C.
* Impaired liver function, as evidenced by serum glutamic-pyruvic transaminase (SGPT) or serum glutamic-oxaloacetic transaminase (SGOT) levels exceeding twice the upper limit of the reference normal range at Visit 1.
* Clinically significant microvascular complications (such as macroalbuminuria, pre-proliferative and proliferative retinopathy), cardiovascular, hepatic, neurological, endocrine, or other systemic conditions, apart from T1D, that may hinder the implementation of the clinical study protocol or the interpretation of study results.
* Scheduled surgery during the study period.
* Mental conditions that affect the subject's ability to comprehend the nature, purpose, and potential consequences of the study.
* Subjects deemed unlikely to adhere to the clinical study protocol, including those with an uncooperative attitude, inability to attend follow-up visits or low likelihood of completing the study.
* Use of an experimental drug or device within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
% time below range (<70 mg/dL) | 12-hour inpatient study
  Percentage of time spent below the target range
Number of Level 1 (<70 mg/dL) and Level 2 (<54 mg/dL) hypoglycemic events | 12-hour inpatient study
  Occurrence of hypoglycemic events during at least 15 min

SECONDARY OUTCOMES:
%time in range (70-180 mg/dL) | 12-hour inpatient study
  Percentage of time spent within target range (70-180 mg/dL)
%time in range (70-140 mg/dL) | 12-hour inpatient study
  Percentage of time spent within target range (70-140 mg/dL)
Time with glucose levels <3.0 mmol/l (54 mg/dl) | 12-hour inpatient study
  Percentage of time spent with glucose levels < 3.0 mmol/l (54 mg/dl)
Coefficient of variation (CV) of CGM values | 12-hour inpatient study
  Glycemic variability
%time >180 mg/dL | 12-hour inpatient study
  Percentage of time spent above 180 mg/dL
%time > 250 mg/dL | 12-hour inpatient study
  Percentage of time spent above 250 mg/dL
Average glucose | 12-hour inpatient study
  Average of sensor glucose levels (mg/dL)
Standard deviation | 12-hour inpatient study
  Standard deviation of sensor glucose levels
Total insulin | 12-hour inpatient study
  Total insulin administered during the inpatient study
Total glucagon | 12-hour inpatient study
  Total glucagon administered during the inpatient study
Number of automatic rescue carbohydrate recommendations | 12-hour inpatient study
  Number of rescue carbohydrate recommendations applied during the inpatient study
Number of glucagon boluses | 12-hour inpatient study
  Number of glucagon boluses administered during the inpatient study
Total number of carbohydrates ingested | 12-hour inpatient study
  Total number of carbohydrates ingested (g) during the inpatient study

CONTACTS AND LOCATIONS:
Overall Officials: F. Javier Ampudia-Blasco, MD PhD, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakshman R, Boughton C, Hovorka R. The changing landscape of automated insulin delivery in the management of type 1 diabetes. Endocr Connect. 2023 Jul 31;12(8):e230132. doi: 10.1530/EC-23-0132. PMID 37289734
- [Background] Eckstein ML, Weilguni B, Tauschmann M, Zimmer RT, Aziz F, Sourij H, Moser O. Time in Range for Closed-Loop Systems versus Standard of Care during Physical Exercise in People with Type 1 Diabetes: A Systematic Review and Meta-Analysis. J Clin Med. 2021 May 31;10(11):2445. doi: 10.3390/jcm10112445. PMID 34072900
- [Background] Brazeau AS, Rabasa-Lhoret R, Strychar I, Mircescu H. Barriers to physical activity among patients with type 1 diabetes. Diabetes Care. 2008 Nov;31(11):2108-9. doi: 10.2337/dc08-0720. Epub 2008 Aug 8. PMID 18689694
- [Background] Paldus B, Morrison D, Lee M, Zaharieva DP, Riddell MC, O'Neal DN. Strengths and Challenges of Closed-Loop Insulin Delivery During Exercise in People With Type 1 Diabetes: Potential Future Directions. J Diabetes Sci Technol. 2023 Jul;17(4):1077-1084. doi: 10.1177/19322968221088327. Epub 2022 Apr 24. PMID 35466723
- [Background] Zaharieva DP, Morrison D, Paldus B, Lal RA, Buckingham BA, O'Neal DN. Practical Aspects and Exercise Safety Benefits of Automated Insulin Delivery Systems in Type 1 Diabetes. Diabetes Spectr. 2023 May;36(2):127-136. doi: 10.2337/dsi22-0018. Epub 2023 May 15. PMID 37193203
- [Background] Wilson LM, Jacobs PG, Castle JR. Role of Glucagon in Automated Insulin Delivery. Endocrinol Metab Clin North Am. 2020 Mar;49(1):179-202. doi: 10.1016/j.ecl.2019.10.008. Epub 2019 Dec 10. PMID 31980117
- [Background] Haidar A. Insulin-and-Glucagon Artificial Pancreas Versus Insulin-Alone Artificial Pancreas: A Short Review. Diabetes Spectr. 2019 Aug;32(3):215-221. doi: 10.2337/ds18-0097. PMID 31462876
- [Background] Taleb N, Emami A, Suppere C, Messier V, Legault L, Ladouceur M, Chiasson JL, Haidar A, Rabasa-Lhoret R. Efficacy of single-hormone and dual-hormone artificial pancreas during continuous and interval exercise in adult patients with type 1 diabetes: randomised controlled crossover trial. Diabetologia. 2016 Dec;59(12):2561-2571. doi: 10.1007/s00125-016-4107-0. Epub 2016 Oct 4. PMID 27704167
- [Background] Laugesen C, Ranjan AG, Schmidt S, Norgaard K. Low-Dose Dasiglucagon Versus Oral Glucose for Prevention of Insulin-Induced Hypoglycemia in People With Type 1 Diabetes: A Phase 2, Randomized, Three-Arm Crossover Study. Diabetes Care. 2022 Jun 2;45(6):1391-1399. doi: 10.2337/dc21-2304. PMID 35475907